CLINICAL TRIAL: NCT03514719
Title: PD-L1 Imaging in Non Small Cell Lung Cancer' (PINNACLE)
Acronym: PINNACLE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MS100070_0167
Record Dates: First submitted 2018-04-20; First posted 2018-05-02 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: 89Zr-avelumab PET; avelumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — avelumab

STUDY DESIGN:
Intervention Model Description: Patients with early stage disease (stage Ia(≥T1b)-IIIa) undergo pre-treatment PET-imaging and 2 cycles of neo-adjuvant avelumab treatment. Followed by surgical resection of the tumor.
  Patients with stage IIIb-IV NSCLC will undergo pre-treatment PET-imaging in only part 1 of the study, and receive avelumab treatment 10mg/kg q2w until disease progression or treatment toxicity
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 89Zr-avelumab PET (Experimental): 89Zr-avelumab injection followed by 89Zr-avelumab PET
  Interventions: Diagnostic Test: 89Zr-avelumab PET; Drug: Avelumab

INTERVENTIONS:
Diagnostic Test: 89Zr-avelumab PET — 89Zr-avelumab injection followed by 89Zr-Avelumab PET scan
  Other Names: ImmunoPET
Drug: Avelumab — Early stage disease (stage Ia (≥T1b tumor)-IIIa: neo-adjuvant avelumab treatment (10mg/kg iv q2w) for a maximum duration of 2 cycles after PET-imaging, followed by surgical resection of the tumor with curative intent
  Stage IIIb-IV disease: systemic treatment with avelumab 10mg/kg iv q2w after PET-imaging

SUMMARY:
In this feasibility study, a zirconium-89 (89Zr)-avelumab positron emission tomography (PET) scan will be performed in 37 patients prior to treatment with avelumab to:

1. assess the tumor and systemic tissue uptake 89Zr-avelumab
2. assess the potential to predict avelumab treatment response

DETAILED DESCRIPTION:
The programmed death 1 (PD1)/ programmed death ligand 1 (PD-L1) pathway plays an important role in regulating the T-cell anti tumor response. Blocking this interaction with the anti PD-L1 monoclonal antibody avelumab is effective in patients with non-small cell lung cancer (NSCLC) resulting in durable disease control rates. Currently, PD-L1 expression as determined by immune histochemistry (IHC) is the best available biomarker for treatment response, but standardized scoring criteria are lacking and the risk for sampling errors exists. Molecular imaging using 89Zr-labeled antibodies may overcome these limitations, enabling the visualization of PD-L1 expression in primary and metastatic tumor lesions and providing information on the in vivo accessibility of the PD-L1 target following intravenous administration.

This study enables PD-L1 PET-imaging with 89Zr-avelumab in patients with:

* early stage NSCLC (stage Ia (≥T1b) -IIIa) followed by 2 cycles of neo-adjuvant avelumab treatment and surgical resection of the tumor.
* advanced stage NSCLC (Stage IIIb-IV) followed by avelumab treatment until disease progression or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥ 18 years, and >50 years in patients with resectable stage Ia (≥T1b tumor) - IIIa NSCLC)
2. Histological or cytologic proven stage IIIb/IV NSCLC or resectable stage Ia (≥T1b tumor) - IIIa NSCLC, where no pathological evaluation of mediastinal lymph nodes by mediastinoscopy is indicated according to the multidisciplinary tumor board
3. ECOG performance score (0-1)
4. At least one lesion with a tumour size ≥ 1 cm
5. Haematologic function: absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L, and haemoglobin ≥ 9 g/dL (may have been transfused)
6. Hepatic function: total bilirubin level ≤ 1.5 × the upper limit of normal (ULN) range and AST and ALT levels ≤ 2.5 × ULN for all subjects or AST and ALT levels ≤ 5 x ULN (for subjects with documented metastatic disease to the liver).
7. Estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method)
8. Highly effective contraception for both male and female subjects throughout the study and for at least after avelumab treatment administration intrinsic factor the risk of conception exists
9. Fit for surgery (for patients with resectable stage Ia-IIIa disease), as assessed by treating thoracic surgeon / anesthesiologists based on sufficient cardiopulmonary status and absence of major contra-indications for surgery according to local guidelines

Exclusion Criteria:

1. Immunosuppressants: "Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (eg, intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication)."
2. Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent: Subjects with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible
3. Prior organ transplantation, including allogeneic stem cell transplantation
4. Infections: active infection requiring systemic therapy
5. HIV/AIDS: known history for testing positive to an HIV test or known acquired immunodeficiency syndrome (AIDS)
6. Hepatitis: hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or confirmatory HCV RNA if anti-HCV antibody screening test positive)
7. Vaccination within 4 weeks of the first dose of avelumab and while on trial is prohibited except for administration of inactivated vaccines
8. Hypersensitivity to study drug: "Known prior severe hypersensitivity reactions to investigational product or any component in its formulations, including known severe hypersensitivity reactions to antibodies (Grade ≥ 3 NCI CTCAE v 4.03)
9. Cardiovascular disease: "Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication."8. Persisting toxicity related to prior therapy of Grade >1 NCI-CTCAE v 4.03; however, alopecia and sensory neuropathy Grade ≤ 2 is acceptable
10. Other persisting toxicities: Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 > 1); however, alopecia, sensory neuropathy Grade

    ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
11. Other severe acute or chronic medical conditions including colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Tumor uptake of 89Zr-Avelumab | 1 year
  Standardized uptake values (SUV) of 89Zr-Avelumab uptake in tumor lesions will be measured

SECONDARY OUTCOMES:
Correlation 89Zr-Avelumab uptake in tumor lesions and PD-L1 expression as determined by immunohistochemistry | 1-2 year
Correlation between 89Zr-Avelumab uptake in tumor lesions and response to (neo)-adjuvant avelumab treatment | 1-2 years
  To assess the potential of PD-L1 PET/CT to image PD-L1 expression in tumor lesions, and predict response to (neo)-adjuvant avelumab treatment in patients with NSCLC
The number of treatment delays in surgical resections | 1-2 years
  In resectable early stage disease (stage Ia (≥T1b) - IIIa)
Asses post-operative complications | 1-2 years
  In resectable early stage disease (stage Ia (≥T1b) - IIIa)

CONTACTS AND LOCATIONS:
Overall Officials: C.M.L. van Herpen, Prof.dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University, Nijmegen, Netherlands